CLINICAL TRIAL: NCT06670651
Title: LinkSymphoKnee (LSK) Total Knee Replacement System Study - Ultra-congruent (UC)
Status: Enrolling by invitation | Type: Observational
Sponsor: LinkBio Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: LB24001-LSKUC
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis (OA) of the Knee; Fracture; Rheumatoid Arthritis
Keywords: primary total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis; Fractures, Bone; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: total knee arthroplasty device — total knee arthroplasty device with ultracongruent bearing surface

SUMMARY:
To collect information about implant performance and patient clinical outcomes in patients undergoing primary total knee arthroplasty with the LinkSymphoKnee total knee replacement system with ultra-congruent tibial bearing surface.

DETAILED DESCRIPTION:
The study will collect outcomes data on up to 600 patients from up to 3 sites using a legally marketed device according to its labeled intended use.

The study will collect:

1. KOOS-JR
2. Knee Society Score (KSS), 2011
3. PROMIS Global Health
4. PROMIS Physical Function
5. PROMIS Pain Interference
6. Surgery Satisfaction
7. Forgotten Joint Score
8. Radiographic findings
9. Revisions.

Radiographic evaluations will be done through postoperative year 2. Other outcomes will be evaluated up to postoperative year 5.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, and skeletally mature; and
* Undergoing a primary TKA for one or both knees using the cemented LinkSymphoKnee knee system as part of the surgeon's standard of care.
* Able to read and understand English (because patient-reported outcome questionnaires are not validated for all potential other languages).

Exclusion Criteria:

* 80 years of age or older,
* Women who are pregnant at the time of surgery,
* History of joint sepsis,
* Bone defect that requires grafting,
* Previous history of bone disease (e.g., severe osteoporosis or osteomalacia) which in the surgeon's opinion is severe enough to compromise device fixation,
* Systemic conditions affecting bone density (e.g., inflammatory arthritis or renal disease) which in the surgeon's opinion are severe enough to compromise device fixation,
* A poorly functioning contralateral total knee replacement or a contralateral revision regardless of function.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking primary total knee arthroplasty from the participating surgeon investigators
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score - Joint Replacement (KOOS-JR) - change from baseline | 1 year postoperative
  Patient-reported outcome measure (PROM) that assesses knee health based on questions about pain, stiffness, function, and daily activities. Minimum score = 0. Maximum score = 100. Higher score means a better outcome.
Revision rate | 5 years postoperative
  Evaluates how often patients require additional surgery to remove or replace the knee arthroplasty device components.

SECONDARY OUTCOMES:
Knee Society Score - change from baseline | postoperative intervals through 5 years
  A rating scale that measures the outcome of a patient's knee replacement surgery by assessing objective and subjective outcomes, including pain, range of motion, stability, walking distance, and ability to climb stairs, and also patient satisfaction and expectations. Minimum score = 0. Maximum score = 100. Higher score means better outcome.
PROMIS Global Health Score - change from baseline | postoperative intervals through 5 years
  PROMIS Global Health measures physical function, pain, fatigue, emotional distress, and social health. The raw score minimum is 7 and maximum is 35. Higher score means better outcome.
Surgery Satisfaction Score | 1 and 5 years postoperative
  Measures a patient's satisfaction with a surgical procedure based on questions about pain control and daily activities. Minimum score is 0. Maximum score is 10. Higher score means better outcome.
Forgotten Joint Score | postoperative intervals through 5 years
  Measures a patient's awareness of their artificial knee joint. Minimum score is 0. Maximum score is 100. Higher score means better outcome.
Knee Society Roentgenographic Evaluation and Scoring System | Through 2 years postoperative
  Evaluates radiographic signs of device stability. 3 zones are assigned to evaluate the patella component. 5-7 zones are assigned to evaluate the tibia and femur components. Radiolucencies are evaluated for size, location, and progression over time. Changes in implant position and/or radiolucencies that are large, continuous, or progressive over time signify possible or impending implant failure.
PROMIS Pain Interference Score - change from baseline | postoperative intervals through 5 years
  The score measures how pain affects a person's life. The raw score minimum is 6 and maximum is 30. A lower score means a better outcome.
PROMIS Physical Function Score - change from baseline | postoperative intervals through 5 years
  The score measures a person's ability to perform activities. The raw score minimum is 11 and maximum is 72.5. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Schwartz, MD, Principal Investigator — Illinois Bone & Joint Institute
Locations (2):
- United States (2):
  - OrthoAlabama Spine & Sports, Birmingham, Alabama
  - Illinois Bone and Joint Institute, Libertyville, Illinois

IPD SHARING:
Plan to Share IPD: No